CLINICAL TRIAL: NCT01077323
Title: A Retrospective Cohort Study of Acute Pancreatitis in Relation to Use of Byetta (Exenatide) and Other Antidiabetic Agents
Brief Title: A Retrospective Cohort Study of Acute Pancreatitis in Relation to Use of Exenatide and Other Antidiabetic Agents
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry); i3 Drug Safety (Other)
Responsible Party: Sponsor
Other Study IDs: BCA406
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes (Treated With Exenatide or Other Oral Antidiabetic Therapies); Healthy Subjects (Treated With no Diabetes Therapies)
Keywords: pancreatitis; exenatide; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pancreatitis | interventions — Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exenatide Initiators
  Interventions: Drug: exenatide
- Other Antidiabetic Drug Initiators
  Interventions: Drug: Other antidiabetic therapies
- Non-Diabetes Cohort
  Interventions: Other: No diabetes therapy

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, dosing according to normal clinical practice
  Other Names: Byetta
  Groups: Exenatide Initiators
Drug: Other antidiabetic therapies — Includes metformin, thiazolidinediones, insulins, sulfonylureas, non-sulfonylurea secretagogues, sitagliptin, and alpha-glucosidase inhibitors; In all cases, dosing according to normal clinical practice
  Groups: Other Antidiabetic Drug Initiators
Other: No diabetes therapy — Subjects not diagnosed with diabetes
  Groups: Non-Diabetes Cohort

SUMMARY:
The purpose of this research was to assess the absolute and relative incidence of acute pancreatitis in persons initiating exenatide compared with persons initiating a different antidiabetic agent, and secondarily, persons without diabetes. This protocol summarizes a retrospective cohort study using eligibility, pharmacy claims, and medical claims data from a large US health plan affiliated with i3 Drug Safety.

DETAILED DESCRIPTION:
Limitations of the study: The results provided below should be interpreted in light of the following limitations:

* Misclassification of acute pancreatitis may have distorted our estimates of absolute and relative IRs. In cases where the degree of misclassification is non-differential with respect to the exposure cohort, as is likely the case in administrative data, the RR would be biased toward the null value, although the magnitude of bias will depend on the amount of misclassification.
* Lack of information on important potential confounders, like obesity and alcohol use, is another limitation of the present analysis. Although we adjusted for propensity scores of exenatide initiation, which included a large number of factors derived from the claims data, it is likely that the present estimates are somewhat inaccurate due to residual confounding.
* Our definition of current use in the time-on-drug analysis, which extended 31 days past the nominal end of the last dispensing of the cohort-defining drug, may be too long in duration and thus misclassify exposure during the relevant etiologic period.
* Additionally, these analyses assume that when pharmacies submit a claim for a medication that patients receive and consume the medication. While it is possible that misclassification of exposure by non-adherence to the medications dispensed occurred, prior work showed that pharmacy claims are valid for ascertaining medication exposure.

ELIGIBILITY:
Inclusion Criteria:

* Exenatide Initiators: The date of the first dispensing of exenatide under which a potential cohort member might qualify will be 1 June 2005, and the latest date will be 31 December 2007. We will note the first initiation of exenatide, and also note subsequent initiation of other antidiabetic drugs. Eligible exenatide initiators will be included in the exenatide initiator cohort on the first eligible dispensing following at least 9 months of continuous health plan enrollment.
* Other Antidiabetic Drug Initiators: The date of the first dispensing of an antidiabetic drug other than exenatide under which a potential cohort member might qualify will be 1 June 2005, and the latest date will be 31 December 2007. We will note the earliest date of other antidiabetic drug dispensings within their cohort membership, and also note subsequent initiation of other antidiabetic drugs. We will choose a subset of this comparator cohort randomly selected to be approximately 9 times larger than the exenatide initiators and will oversample patients receiving certain drugs to the extent necessary to ensure inclusion of at least as many persons initiating these drugs as initiating exenatide. Specifically, oversampling will be performed as needed on initiators of metformin, TZDs, SUs, sitagliptin and insulin glargine to allow for further sub-analysis.
* Exenatide and Other Antidiabetic Drug Initiators: For all patients in these two study cohorts, the date of cohort entry (the date ranged between January 1, 2005 and December 31, 2007) marked the beginning of observation for study outcomes (follow-up). The end of observation for a given patient happened on the earliest of occurrence of likely acute pancreatitis, end of the study period (March 31, 2008), or disenrollment from the health plan.
* Non-Diabetes Cohort: A third cohort will consist of randomly-selected Ingenix Research Data Mart members who have no claim associated with a diabetes diagnosis or antidiabetic drug dispensing in the baseline continuous enrollment period. This cohort will enter as of the later of 1 June 2005 or completion of 9 months continuous baseline enrollment and will provide follow-up through end of enrollment or 31 March 2008, or the receipt of an antidiabetic drug dispensing or diabetes diagnosis, at which point they may enter one of the other exposure cohorts.

Exclusion Criteria:

* The 3 cohorts (exenatide initiators, other antidiabetic initiators, and those without diabetes) will be subject to minimal exclusions in order to observe acute pancreatitis across a wide spectrum of patient characteristics. We will apply a baseline enrollment requirement of 9 months prior to cohort entry so that the first day of follow-up (on which acute pancreatitis could occur) will be characterized with the same level of detail (based on 9 months of preceding health insurance claims) as any other day during the study.
* Consistent with the principle of minimal exclusions, we will only exclude from the cohorts people who have baseline claims associated with pancreatitis (in the 9-month period preceding cohort entry) as these people either had pre-existing pancreatitis or had a pre-existing suspicion of pancreatitis. We will not exclude persons with a type I diabetes diagnosis as we intend to observe the spectrum of clinical practice with respect to antidiabetic drug initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study utilized medical claims data from a large US health plan affiliated with i3 Drug Safety. The individuals covered by this health plan are geographically diverse across the United States. The health plan provides fully insured coverage for physician, hospital and prescription drug services. The providers of these services submit their claims for payment directly to the health plan. i3 Drug Safety uses de-identified data derived from these claims daily for a wide range of safety, utilization, and economic analyses.
Sampling Method: Non-Probability Sample
Enrollment: 363766 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Research and Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (1):
- Research Site, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Initiators: Exenatide initiators were persons with a pharmacy claim associated with a dispensing of exenatide preceded by 9 months of continuous enrollment in the underlying health insurance plan without an exenatide dispensing. Patients eligible for both the exenatide cohort and the other antidiabetic drug medication cohort were preferentially entered into the former.
- Other Antidiabetic Drug (OADs) Initiators: Initiators of other antidiabetic medications were persons with a pharmacy claim associated with a dispensing of one of the following drugs preceded by 9 months of continuous enrollment in the underlying health insurance program without a dispensing of the same medication: sulfonylureas (e.g. glyburide); metformin; TZDs (e.g. rosiglitazone); insulins (e.g. insulin glargine); sitagliptin; pramlintide; non-sulfonylurea secretagogues (e.g. repaglinide); α-glucosidase inhibitors (e.g. miglitol).
- Non-Diabetes Cohort: The Non-Diabetes Cohort was composed of persons who had 9 months of continuous enrollment in the underlying health insurance program prior to their assigned index dates and no claims associated with a diagnosis of diabetes, no dispensing of a diabetes drug, and no diagnosis of pancreatic disease in the baseline period.
Period: Overall Study
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Started | 37097 (STARTED = Number of subjects considered for inclusion in this cohort.) | 620799 (STARTED = Number of subjects considered for inclusion in this cohort.) | 12015600 (STARTED = Number of subjects considered for inclusion in this cohort.)
Completed | 25719 (COMPLETED = Group of subjects for whom data in outcome measures is presented.) | 234536 (COMPLETED = Group of subjects for whom data in outcome measures is presented.) | 103511 (COMPLETED = Group of subjects for whom data in outcome measures is presented.)
Not Completed | 11378 | 386263 | 11912089
Not completed — <9 months enroll before drug dispensed | 11226 | 263954 | 11655523
Not completed — Dispensing of drug in baseline period | 0 | 120229 | 256446
Not completed — Baseline diagnosis of pancreatic disease | 152 | 2080 | 120

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort | Total
Number analyzed (Participants) | 25719 | 234536 | 103511 | 363766
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 2982 | 24963 | 27999
  Between 18 and 65 years | 23496 | 202317 | 73622 | 299435
  >=65 years | 2169 | 29237 | 4926 | 36332
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14381 | 114960 | 52444 | 181785
  Male | 11338 | 119576 | 51067 | 181981
Has a History of Congestive Heart Failure [Number; unit: participants] — Has a History of Congestive Heart Failure
  participants | 820 | 8227 | 315 | 9362
Has a History of Hyperlipidemia [Number; unit: participants] — Has a History of Hyperlipidemia
  participants | 19741 | 127384 | 13178 | 160303
Has a History of Hypertension [Number; unit: participants] — Has a History of Hypertension
  participants | 16336 | 114593 | 10121 | 141050
Has a History of Ischemic Heart Disease [Number; unit: participants] — Has a History of Ischemic Heart Disease
  participants | 3228 | 24900 | 1775 | 29903
Has a History of Myocardial Infarction [Number; unit: participants] — Has a History of Myocardial Infarction
  participants | 301 | 3951 | 193 | 4445
Has a History of Obesity [Number; unit: participants] — Has a History of Obesity
  participants | 4107 | 18933 | 1230 | 24270
Has a History of Peripheral Neuropathy [Number; unit: participants] — Has a History of Peripheral Neuropathy
  participants | 2456 | 9581 | 11 | 12048
Has a History of Renal Impairment/Dialysis [Number; unit: participants] — Has a History of Renal Impairment/Dialysis
  participants | 961 | 8257 | 312 | 9530
Has a History of Retinopathy [Number; unit: participants] — Has a History of Retinopathy
  participants | 1279 | 6693 | 76 | 8048
Has a History of Stroke/Transient Ischemic Attack [Number; unit: participants] — Has a History of Stroke/Transient Ischemic Attack
  participants | 423 | 5088 | 336 | 5847
Has a History of Type 1 Diabetes [Number; unit: participants] — Has a History of Type 1 Diabetes
  participants | 2794 | 19368 | 0 | 22162
Has a History of Type 2 Diabetes [Number; unit: participants] — Has a History of Type 2 Diabetes
  participants | 21709 | 138218 | 0 | 159927

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates Per 100,000 Person-Years of Likely Acute Pancreatitis (During "Current Use" Period) - Time on Drug Analysis
Description: Crude time-on-drug incidence rate per 100,000 person-years of likely acute pancreatitis in initiators of exenatide, initiators of other antidiabetic drugs and the non-diabetes cohort. Analysis period is "current use" period, described as "time during current day's supply plus 31 days."
Time Frame: 43 months
Population: Time on Drug Analysis
Measure: Number (95% Confidence Interval); unit: Cases per 100,000 person-years
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Number analyzed (Participants) | 25719 | 234536 | 103511
Cases per 100,000 person-years | 219.7 [155.5 to 301.6] | 226.7 [205.4 to 249.6] | 56.2 [43.7 to 71.1]
Statistical Analysis 1: Comparison: Exenatide Initiators vs Other Antidiabetic Drug (OADs) Initiators; Test type: Superiority or Other; Adjusted Rate Ratio (ARR) = 0.87, 95% CI 2-sided [0.59 to 1.28] — ARR equals adjusted incidence rate of acute pancreatitis in exenatide cohort divided by adjusted incidence of acute pancreatitis in OAD cohort. Adjusted incidence rates were calculated using a Poisson regression model adjusted for propensity score

2. Secondary Outcome: Incidence Rates Per 100,000 Person-Years of Likely Acute Pancreatitis Among Initiators of Exenatide, Diabetics Initiating Other Antidiabetic Drugs, and the Non-diabetes Cohort - Intent to Treat Analysis
Description: Crude intent-to-treat incidence rate per 100,000 person-years of likely acute pancreatitis in initiators of exenatide, initiators of other antidiabetic drugs and the non-diabetes cohort.
Time Frame: 43 months
Population: Intent to Treat Analysis
Measure: Number (95% Confidence Interval); unit: Cases per 100,000 person-years
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Number analyzed (Participants) | 25719 | 234536 | 103511
Cases per 100,000 person-years | 272.7 [215.6 to 340.4] | 227.6 [209.4 to 246.9] | 56.2 [43.7 to 71.1]
Statistical Analysis 1: Comparison: Exenatide Initiators vs Other Antidiabetic Drug (OADs) Initiators; Test type: Superiority or Other; Adjusted Rate Ratio (ARR) = 1.1, 95% CI 2-sided [0.8 to 1.5] — ARR equals adjusted incidence rate of acute pancreatitis in exenatide cohort divided by adjusted incidence of acute pancreatitis in OAD cohort.Rate ratios adjusted for propensity score of exenatide initiation using Cox Proportional Hazards Regression

3. Primary Outcome: Incidence Rates Per 100,000 Person-Years of Likely Acute Pancreatitis (Among "Recent Use" Period) - Time on Drug Analysis
Description: Crude time-on-drug incidence rate per 100,000 person-years of likely acute pancreatitis in initiators of exenatide, initiators of other antidiabetic drugs and the non-diabetes cohort. Analysis period is the "recent use" period, described as "time following current use plus an additional 31 days excluding subsequent current use."
Time Frame: 43 months
Population: Time on Drug Analysis
Measure: Number (95% Confidence Interval); unit: Cases per 100,000 person-years
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Number analyzed (Participants) | 25719 | 234536 | 103511
Cases per 100,000 person-years | 321.4 [117.9 to 699.5] | 325.5 [243.8 to 425.7] | 56.2 [43.7 to 71.1]
Statistical Analysis 1: Comparison: Exenatide Initiators vs Other Antidiabetic Drug (OADs) Initiators; Test type: Superiority or Other; Adjusted Rate Ratio (ARR) = 0.87, 95% CI 2-sided [0.36 to 2.09] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Incidence Rates Per 100,000 Person-Years of Likely Acute Pancreatitis (During "Past Use" Period) - Time on Drug Analysis
Description: Crude time-on-drug incidence rate per 100,000 person-years of likely acute pancreatitis in initiators of exenatide, initiators of other antidiabetic drugs and the non-diabetes cohort. Analysis period is "past use" period, described as "time following recent use excluding subsequent current or recent use."
Time Frame: 43 months
Population: Time on Drug Analysis
Measure: Number (95% Confidence Interval); unit: Cases per 100,000 person-years
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Number analyzed (Participants) | 25719 | 234536 | 103511
Cases per 100,000 person-years | 354.5 [245.5 to 495.4] | 218.1 [183.0 to 258.0] | 56.2 [43.7 to 71.1]
Statistical Analysis 1: Comparison: Exenatide Initiators vs Other Antidiabetic Drug (OADs) Initiators; Test type: Superiority or Other; Adjusted Rate Ratio (ARR) = 1.39, 95% CI 2-sided [0.86 to 2.25] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: SERIOUS ADVERSE EVENTS AND ADVERSE EVENTS NOT APPLICABLE (please see additional description below).
Description: This study was an epidemiological, retrospective study specifically looking at the incidence of acute pancreatitis in exenatide initiators, OAD initiators, and a non-diabetes cohort. Adverse events, other than pancreatitis, were not evaluated in this study. All data was deidentified and the severity of acute pancreatitis disease was not evaluated.
Arm/Group | Exenatide Initiators | Other Antidiabetic Drug (OADs) Initiators | Non-Diabetes Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less